CLINICAL TRIAL: NCT01066702
Title: A Randomized Comparison of NeoCart to Microfracture for the Repair of Articular Cartilage Injuries in the Knee
Brief Title: Confirmatory Study of NeoCart in Knee Cartilage Repair
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: company dissolution
Sponsor: Histogenics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8-01
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2018-12

CONDITIONS: Articular Cartilage Defects in the Knee Joint
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NeoCart (Experimental): Autologous cartilagenous tissue implant
  Interventions: Biological: NeoCart
- Microfracture (Active Comparator): surgical intervention
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Biological: NeoCart — implantation of an cartilagenous tissue implant derived from the patients own cells.
  Arms: NeoCart
Procedure: Microfracture — holes are created in bone at the base of the defect bed to encourage growth of tissue within the defect bed.
  Arms: Microfracture

SUMMARY:
This confirmatory study is a prospective randomized trial comparing the efficacy and safety of an autologous chondrocyte tissue implant (NeoCart) to the surgical intervention microfracture in the treatment of cartilage defects in the knee.

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 years old
* symptomatic articular cartilage lesion of the femur and/or trochlea

Exclusion Criteria:

* prior surgical intervention other than debridement
* arthritis
* clinically significant or symptomatic vascular or neurologic disorder of the lower extremities

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 245 (Actual)
Dates: Start 2010-05; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
The change of physical functioning and pain as assessed by patient reported outcome measures (Knee injury and Osteoarthritis Outcome Score (KOOS), International Knee Documentation Committee (IKDC) score) | one year

SECONDARY OUTCOMES:
Repair cartilage structure as measured by magnetic resonance imaging (MRI) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Belschner, Study Director — Histogenics Corporation
Locations (31):
- United States (29):
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Grossmont Orthopedic Medical Group, La Mesa, California
  - Orthopaedic Specialty Institute/Newport Orthopedic Institute (OSI/NOI), Orange, California
  - UCSF Mission Bay Orthopaedic Institute, San Francisco, California
  - Southern California Orthopedic Research and Education, Van Nuys, California
  - Colorado University Boulder, Boulder, Colorado
  - Steadman Hawkins Clinic - Denver, Denver, Colorado
  - Shrock Clinical Research, Fort Lauderdale, Florida
  - Jewett Orthopaedic Clinic, Orlando, Florida
  - Optim Healthcare, Savannah, Georgia
  - St. Lukes Medical Center, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - OrthoIndy, Greenwood, Indiana
  - Ochsner Clinic Sports Medicine, New Orleans, Louisiana
  - Orthopaedic Associates, Portland, Maine
  - Harvard Vanguard Medical Associates, West Roxbury, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - TRIA Orthopaedic Center, Bloomington, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Alpine Orthopedics & Sports Medicine, Bozeman, Montana
  - University of New Mexico, Albuquerque, New Mexico
  - Hospital for Special Surgery, New York, New York
  - Duke Sports Medicine, Durham, North Carolina
  - Ohio State University - Department of Sports Medicine, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The San Antonio Orthopaedic Group (TSAOG), San Antonio, Texas
  - The Orthopedic Specialty Hospital, Murray, Utah
  - University of Washington, Seattle, Washington
- Canada (2):
  - Simon Fraser Orthopaedic Fund, New Westminster, British Columbia
  - Fowler Kennedy Sports Medicine Clinic, London, Ontario

REFERENCES:
- [Background] Crawford DC, DeBerardino TM, Williams RJ 3rd. NeoCart, an autologous cartilage tissue implant, compared with microfracture for treatment of distal femoral cartilage lesions: an FDA phase-II prospective, randomized clinical trial after two years. J Bone Joint Surg Am. 2012 Jun 6;94(11):979-89. doi: 10.2106/JBJS.K.00533. PMID 22637204
- [Background] Crawford DC, Heveran CM, Cannon WD Jr, Foo LF, Potter HG. An autologous cartilage tissue implant NeoCart for treatment of grade III chondral injury to the distal femur: prospective clinical safety trial at 2 years. Am J Sports Med. 2009 Jul;37(7):1334-43. doi: 10.1177/0363546509333011. Epub 2009 May 15. PMID 19448048
- See also: Histogenics WebSite — http://www.histogenics.com